CLINICAL TRIAL: NCT07027215
Title: Impact of Augmented Sensory Feedback on Motor Control and Risk of Falling in Cancer-Related Neuropathic Patients"
Brief Title: Augmented Sensory in Cancer-Related Neuropathic Patients"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University, Jordan (Other)
Responsible Party: Principal Investigator, Abeer Abdrabo, Lecture of physical Therapy, Department of Neuromuscular Disorder, Faculty for Physical Therapy, Cairo University, Cairo, Egypt, Isra University, Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Augmented Sensory Feedback
Record Dates: First submitted 2025-06-07; First posted 2025-06-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group 20 Patients" (Active Comparator): Cancer-Related Neuropathic Patients"
  Interventions: Combination Product: selected physical therapy program as arm excercises
- study group 20 Patients" (Active Comparator): Cancer-Related Neuropathic Patients"
  Interventions: Combination Product: Gradual Intermittent pneumatic compression therapy (IPC),Balance excercises.PNF technique

INTERVENTIONS:
Combination Product: Gradual Intermittent pneumatic compression therapy (IPC),Balance excercises.PNF technique — PNF technique
  Other Names: Balance Exercises
  Arms: study group 20 Patients"
Combination Product: selected physical therapy program as arm excercises — selected physical therapy program only. The program consisted of (core exercises, AROM exercises, and stretching exercises for LL for 18 sessions every other day, over 6 weeks
  Arms: control group 20 Patients"

SUMMARY:
this research studied the effect of augmented sensory feedback program on motor control and risk of falling in patient with CIPN.

DETAILED DESCRIPTION:
Design: A randomized control trial was conducted to investigate the impact of augmented sensory feedback paradigm on motor control and risk of falling in patient with Chemotherapy-induced peripheral neuropathy. Data were collected pre and post treatment from out-patient clinic of the Faculty of Medicine and Faculty of Physical Therapy South Valley University, between January 2023and March 2024. The study was approved by the ethical committee of the Faculty of Physical Therapy, South Vally University, Egypt. The study protocol was explained in detail to every patient and signed written consent was obtained before participation.

Participants: forty female patients with CIPN were recruited from out-patient clinic of the Faculty of Medicine and Faculty of Physical Therapy South Valley University, between January 2023and March 2024.

ELIGIBILITY:
Inclusion Criteria:

* Forty female with age from 35-60 years
* clinically diagnosed with CIPN after recovery from stage I or II breast cancer
* The strength at the toes, ankles, knees, and hips, as determined by manual muscle tests, of at least 3/5.
* The patients can walk independently with or without any assistive devices.

Exclusion Criteria:

* Patients with a history of hereditary peripheral neuropathy
* Diseases that may contribute to peripheral nerve damage, such as diabetes or renal insufficiency, alcohol abuse, HIV, and vasculitis.
* Patient who had central or peripheral neurologic disease, brain or spinal cord metastases
* Orthopedic problems influencing gait, or foot ulcer at the moment of intake.
* Patients with vestibular or neurological problems influencing gait parameters
* Subjects who had participated in regular exercise, as defined as 150 min of light-to-moderate intensity exercise per week over the past year, were excluded from this trial.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients
Enrollment: 40 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
improvement of balance which was assessed by fall risk scale | one and half month
  improvement in feet sensitivity and motor control and risk of falling in both groups in favor of the study group.
Stability measures | one and half month
  postural stability was measured using a Biodex Balance System SD (950-440 with version 4.X software)
Sensory feedback | one and half month
  Sensory feedback was assessed by using Semmes-Weinstein monofilament (SWM)

CONTACTS AND LOCATIONS:
Overall Officials: Abeer A Mohammed, PhD, Principal Investigator — Isra university. Amman.jordan
Locations (1):
- Faculty of Physical Therapy South Valley University, Luxor, Qena Governorate, Egypt

REFERENCES:
- [Result] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Result] Schneberger S. "Prolife" perinatologist. N Engl J Med. 1992 Sep 10;327(11):812; author reply 813-4. No abstract available. PMID 1501662
- [Result] Sienko KH, Seidler RD, Carender WJ, Goodworth AD, Whitney SL, Peterka RJ. Potential Mechanisms of Sensory Augmentation Systems on Human Balance Control. Front Neurol. 2018 Nov 12;9:944. doi: 10.3389/fneur.2018.00944. eCollection 2018. PMID 30483209